CLINICAL TRIAL: NCT01540071
Title: A Phase II Trial of NRX 194204 in Castration- and Taxane-Resistant Prostate Cancer
Brief Title: Trial of NRX 194204 in Castration- and Taxane-Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Io Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4204-202-2011
Record Dates: First submitted 2011-11-13; First posted 2012-02-28 (Estimated); Results first posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-04

CONDITIONS: Castration Resistant Prostate Cancer
Keywords: HRPC (Hormone refractory prostate cancer); Androgen independent prostate cancer; CRPC (Castration and Taxane Resistant Prostate Cancer)
MeSH Terms: interventions — AGN 194204

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NRX 194204 (Experimental): This was a single arm open-label study. All patients enrolled received 20 mg of IRX4204 per day orally, for six months, or longer if the patient had disease stabilization and was tolerating the experimental treatment.
  Interventions: Drug: NRX 194204

INTERVENTIONS:
Drug: NRX 194204 — NRX 194204 is an oblong, soft, gelatin capsule and will be taken once a day
  Other Names: Rexinoid

SUMMARY:
This study is to evaluate the benefits of investigational drug, NRX 194204 in slowing down/stopping/reversing progression of the castration resistant and taxane resistant prostate cancer.

DETAILED DESCRIPTION:
Numerous studies in pre-clinical models and in human clinical trials have clearly established the potential for the use of rexinoids in the treatment and prevention of cancer. NRX 194204, a second generation rexinoid, is a highly potent and specific activator of RXRs (retinoid X receptors). Because NRX 194204 is significantly more selective for the RXRs relative to the RARs (retinoic acid receptors) than a first generation approved drug, it is associated with fewer adverse events in clinical use. This study seeks to investigate NRX 194204 monotherapy in patients with castration- and taxane- resistant prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed prostate cancer
* Documented progression on at least one prior hormone treatment, AND at least one taxane based chemotherapy regimen, or patient's refusal of chemotherapy treatment
* Male, Age > 18 years
* ECOG (Eastern Cooperative Oncology Group) performance score of 0-2
* Adequate bone marrow, renal and hepatic function
* Men of childbearing potential must consent to use barrier contraception while on treatment and for 90 days thereafter

Exclusion Criteria:

* Prior treatment with NRX 194204 or bexarotene (Targretin)
* Presence of parenchymal brain metastases
* History of prior malignancy within the past 5 years with the exception of curatively treated basal cell or squamous cell carcinoma of the skin or superficial bladder or other stage I or stage II cancer in complete remission for at least 12 months
* Patients with a history of unstable or newly diagnosed angina pectoris, documented history of current serious arrhythmia or congestive heart failure or myocardial infarction within 6 months of enrollment
* Known HIV or hepatitis B or C infection
* Life expectancy < 3 months
* Patients with any history of thyroid disease, pituitary disease or treatment with thyroid replacement hormone
* Patients with a history of pancreatitis or at significant risk of developing pancreatitis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lalita Pandit, MD, Principal Investigator — Lalita Pandit, MD
Locations (1):
- Lalita Pandit, MD, Fountain Valley, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 38 patients were recruited
Groups:
- NRX 194204: NRX 194204 capsules, 20 mg PO once per day
Period: Overall Study
Arm/Group | NRX 194204
Started | 38
Completed | 38
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- NRX 194204: NRX 194204, 20 mg orally once per day
Arm/Group | NRX 194204
Number analyzed (Participants) | 38
Age, Continuous [Mean (Full Range); unit: years] | 71.6 [48 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit of NRX 194204 in Men With Castration- and Taxane-resistant Metastatic Prostate Cancer
Description: Clinical benefit will be defined as either non-progression at 8 weeks or radiologic and/or PSA response at any time point with no dose limiting toxicity (DLT) or other toxicity requiring termination of treatment.
Time Frame: participants will be followed for the duration of treatment and follow up, which is up to 2.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | NRX 194204
Number analyzed (Participants) | 38
Participants | 19

2. Secondary Outcome: Overall Survival
Description: Overall Survival [Time Frame: participants will be followed for the duration of treatment and follow up, which is up to 2.5 years]
Time Frame: participants will be followed for the duration of treatment and follow up, which is up to 2.5 years
Measure: Mean (Full Range); unit: days
Groups:
- NRX 194204: This was a single arm open-label study. All patients enrolled and treated received 20 mg of IRX4204 per day orally, for six months, or longer if the patient had disease stabilization and was tolerating the experimental treatment.
Arm/Group | NRX 194204
Number analyzed (Participants) | 38
days | 312 [38 to 933]

3. Secondary Outcome: Time to Disease Progression
Description: Time to Disease Progression was evaluated according to the Response Evaluation Criteria in Solid Tumors (RECIST) guidelines, version 1.1. Progression was defined as at least a 20% relative increase and an absolute increase of at least 5mm; or appearance of new lesions.
Time Frame: participants were to be followed for the duration of treatment and follow up; for up to 2.5 years from baseline
Measure: Mean (Full Range); unit: days
Arm/Group | NRX 194204
Number analyzed (Participants) | 36
days | 105 [21 to 540]

4. Secondary Outcome: Number of Grade 3 and Higher Adverse Events Deemed at Least Possibly Related to NRX 194204
Description: Number of Grade 3 and higher Adverse Events deemed at least possibly related to NRX 194204
Time Frame: participants will be followed for the duration of treatment and follow up, which is up to 2.5 years
Measure: Number; unit: events
Arm/Group | NRX 194204
Number analyzed (Participants) | 38
events | 23

5. Secondary Outcome: PSA Response Rate
Description: Prostate specific Antigen (PSA) response rate based on 50% reduction from baseline PSA
Time Frame: participants will be followed for the duration of treatment and follow up, which is up to 2.5 years
Measure: Number; unit: participants
Arm/Group | NRX 194204
Number analyzed (Participants) | 36
participants
  partial response | 1
  stable disease | 6
  progressive disease | 29

ADVERSE EVENTS:
Time Frame: Adverse events were collected as long as each individual patient was receiving study drug, and were further followed for each individual patient for up to a maximum of 2.5 years, or until they were lost to follow-up, or died.
Arm/Group | NRX 194204
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 13/38
Other Adverse Events (participants affected / at risk) | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NRX 194204 (N=38)
Elevated PT (Blood and lymphatic system disorders) | 1 (1)
Elevated INR (Blood and lymphatic system disorders) | 1 (1)
Elevated PTT (Blood and lymphatic system disorders) | 1 (1)
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 1 (1)
Confusion (Nervous system disorders) | 2 (2)
Hallucinations (Nervous system disorders) | 1 (1)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Probable Upper Gastrointestinal Bleed (Gastrointestinal disorders) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rectal Bleeding (Renal and urinary disorders) | 1 (1)
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Congestive Heart Failure (Cardiac disorders) | 2 (2)
Viral Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Enterococcus Bacteremia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NRX 194204 (N=38)
Hypothyroidism (Endocrine disorders) | 12 (12)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 15 (15)
Fatigue (Metabolism and nutrition disorders) | 13 (13)
Anorexia (Metabolism and nutrition disorders) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 6 (6)
Leucocytopenia (Blood and lymphatic system disorders) | 6 (6)
Urinary Tract Infection (Renal and urinary disorders) | 2 (2)
Increase Alkaline Phosphatase (Hepatobiliary disorders) | 2 (2)
Hypercholesterolemia (Metabolism and nutrition disorders) | 5 (5)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No